CLINICAL TRIAL: NCT06117423
Title: Investigating the Safety, Feasibility, and Optimal Dose of Fluorescently Labeled Adalimumab-680LT for Visualizing Drug Targeting in Inflammatory Bowel Diseases
Brief Title: Fluorescence Imaging of Adalimumab-680LT in Inflammatory Bowel Disease
Acronym: GUIDE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. W.B. Nagengast, MD, prof. dr., University Medical Center Groningen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 18146; 2023-508391-11-00 (Other: CTIS)
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: Fluorescence Molecular Endoscopy; Inflammatory Bowel Disease; Adalimumab-680LT
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No administration of adalimumab-680LT (Other): Patients did not receive adalimumab-680LT, but underwent a Fluorescence Molecular Imaging procedure to serve as a control group and compare results with patients receiving the tracer
  Interventions: Other: Control
- 4.5 mg adalimumab-680LT (Experimental): Patients received 4.5 mg adalimumab-680LT and underwent a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Adalimumab-680LT
- 15 mg adalimumab-680LT (Experimental): Patients received 15 mg adalimumab-680LT and underwent a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Adalimumab-680LT
- 25 mg adalimumab-680LT (Experimental): Patients received 25 mg adalimumab-680LT and underwent a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Adalimumab-680LT
- >14 weeks of adalimumab therapy + optimal dose adalimumab-680LT (Experimental): Patients who received the optimal dose during the first Fluorescence Molecular Imaging procedure are invited for a second procedure after at least 14 weeks of adalimumab therapy. They will receive the optimal dose adalimumab-680LT and will undergo another Fluorescence Molecular Imaging procedure
  Interventions: Drug: Adalimumab-680LT

INTERVENTIONS:
Drug: Adalimumab-680LT — First, adalimumab-680LT was administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure was performed to enable the visualisation and detection of fluorescence signals.
  Arms: 15 mg adalimumab-680LT; 25 mg adalimumab-680LT; 4.5 mg adalimumab-680LT; >14 weeks of adalimumab therapy + optimal dose adalimumab-680LT
Other: Control — Fluorescence Molecular Imaging was performed to enable the visualisation and detection of fluorescence signals.
  Arms: No administration of adalimumab-680LT

SUMMARY:
Crohn's Disease (CD) and Ulcerative Colitis (UC) are chronic inflammatory bowel diseases (IBD). Adalimumab is a human monoclonal antibody against TNF-alpha, a pro-inflammatory cytokine that mediates the inflammatory response in IBD upon binding to the TNF receptors. Primary non-response to adalimumab is high in both CD and UC. Currently, there are no predictors of response to adalimumab and the actual mechanism of action has not yet been elucidated. To gain better understanding of the drug targeting of adalimumab in IBD, the University Medical Center Groningen (UMCG) developed fluorescently labeled adalimumab (adalimumab-680LT). This study aims to assess the safety and the optimal dose of adalimumab-680LT to visualize and potentially quantify the local drug concentration and predict treatment response in IBD patients using in vivo and ex vivo fluorescence molecular imaging (FMI).

ELIGIBILITY:
Inclusion Criteria:

* Established IBD diagnosis (UC or CD)
* Active disease (clinically defined as at least mild activity using dedicated scoring indices and biochemically defined by a fecal calprotectin > 60 µg/g, measured within the last 6 weeks before inclusion)
* Patients must be eligible for adalimumab therapy
* Clinical indication for an endoscopic procedure
* Age: 18 years or older
* Written informed consent
* For female patients of premenopausal age with intact reproductive organs or who are less than 2 years postmenopausal, a negative pregnancy test must be available.

Exclusion Criteria:

* Pregnancy or breast feeding
* Female patient of premenopausal age who does not use any reliable form of contraception at the time of adalimumab-680LT administration and the following 10 weeks.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Prior anti-TNF therapy in the last 6 weeks before inclusion
* Active extra gastrointestinal manifestations of Crohn's disease
* Previous treatment with adalimumab and detectable anti-adalimumab antibodies levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of adalimumab-680LT in IBD | Until 24 hours after administration
  Evaluating possible (severe) adverse events (SAE & AEs)
Blood pressure | Five minutes before, and five and sixty minutes after tracer administration
  Millimeters of mercure (mmHg)
Heart rate | Five minutes before, and five and sixty minutes after tracer administration
  Beats per minute
Temperature | Five minutes before, and five and sixty minutes after tracer administration
  Degrees Celsius
Investigate the feasibility of using FME to detect adalimumab-680LT signals | 12 months
  Evaluating the performance of FME for detecting adalimumab-680LT signals. This evaluation will be based on a visual evaluation during FME (visible signal yes/no), TBR and CNR calculations and MDSFR/SFF measurements.
Investigate the feasibility of using ex vivo FMI to detect adalimumab-680LT | 12 months
  Evaluating the performance of ex vivo FMI for detecting adalimumab-680LT signals. This evaluation will be based on mean fluorescence intensities (MFIs) of biopsies and fluorescence/light sheet microscopy.
Determining the optimal imaging dose of adalimumab-680LT | 12 months
  The optimal dose will be based on the adalimumab-680LT signals during FME and ex vivo FMI

SECONDARY OUTCOMES:
Investigate a potential correlation of in vivo fluorescence signal intensities and target saturation to clinical response/remission after 14 weeks of adalimumab therapy regimen in patients with IBD | 12 months
  Evaluation of the potential correlation in vivo will be based on in vivo fluorescence images and the MDSFR/SFF measurements before and after at least 14 weeks of adalimumab treatment
Investigate a potential correlation of ex vivo fluorescence signal intensities and target saturation to clinical response/remission after 14 weeks of adalimumab therapy regimen in patients with IBD | 12 months
  Evaluation of the potential correlation ex vivo will be based on MFIs of biopsies, fluorescence microscopy results, and tracer concentrations inside biopsies before and after at least 14 weeks of adalimumab treatment
Quantify the fluorescence signals of the tracer in vivo by using single-fiber reflectance/single-fiber fluorescence (MDSFR/SFF) spectroscopy and correlate these measurements to tracer dose, in vivo fluorescence intensities and inflammation severity | 12 months
  Quantification of MDSFR/SFF measurements in inflamed tissue compared to measurements in non-inflamed tissue. Positive correlation between MDSFR/SFF measurements and dose/inflammation severity?
To correlate ex vivo fluorescence signals to inflammation severity and tracer dose based on histopathological examination inside the obtained biopsies | 12 months
  Histologically ascertained tissue types (qualitative):
  Normal (non-inflamed) ileal, colon and rectal tissue Inflamed ileum, colon and rectum tissue Random ''high-fluorescent'' tissue Random ''Non-fluorescent'' tissue
To assess tracer stability, tracer distribution and tracer concentration, and to identify the composition of immune cells ex vivo to learn more about adalimumab mucosal target cells | 12 months
  Fluorescence (confocal) microscopy with additional use of immune panels and spatial transcriptomics analysis (before and after at least 14 weeks of adalimumab treatment). Measurements of the adalimumab-680LT concentration by light-sheet microscopy after tissue clearing, insights in adalimumab-target cells and presence of immune cells inside the biopsies and blood samples by flow cytometry and assessment of tracer stability by Western Blot

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No